CLINICAL TRIAL: NCT06733506
Title: A Pilot Study to Evaluate the Acceptability and Feasibility of Skin Swabbing With Chlorhexidine Gluconate to Prevent Skin And Soft Tissue Infections Among People Who Inject Drugs
Brief Title: A Pilot Study to Evaluate Skin Swabbing With Chlorhexidine to Prevent Skin And Soft Tissue Infections Among People Who Inject Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gabriel John Culbert (Other)
Responsible Party: Sponsor-Investigator, Gabriel John Culbert, Associate Professor, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-0488
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder; Injection Drug Use; Skin and Soft Tissue Infections (SSTIs)
Keywords: opioid use disorder; injection drug use; skin and soft tissue infection; chlorhexidine; people who inject drugs
MeSH Terms: conditions — Opioid-Related Disorders; Soft Tissue Infections | interventions — chlorhexidine gluconate; 2-Propanol; Illicit Drugs

STUDY DESIGN:
Intervention Model Description: All participants received a brief safer-injection training (Intervention A), which consisted of a one-to-one private discussion with a healthcare provider lasting ~5-10 minutes to encourage skin swabbing prior to drug injection. In addition, participants randomized to a Chlorhexidine swab group received a 2-week supply of chlorhexidine swabs which they were instructed to use for 2 weeks, while those randomized to a usual care condition were supplied with a 2-week supply of standard care isopropyl alcohol swabs.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chlorhexidine Swabs (Experimental): Participants randomized to the experimental condition received a 2-week supply of chlorhexidine gluconate pre-saturated, single-use swabs that they were instructed to use for cleaning their skin prior to injecting for the next 2 weeks.
  Interventions: Drug: Chlorhexidine gluconate; Behavioral: Skin Prep Before Injecting Recreational/Street Drugs
- Usual Care (Active Comparator): Participants randomized to a usual care condition received a 2-week supply of isopropyl alcohol swabs that that they were instructed to use for the next 2 weeks to clean their skin prior to injecting.
  Interventions: Drug: Isopropyl Alcohol 70% Topical Application Solution; Behavioral: Skin Prep Before Injecting Recreational/Street Drugs

INTERVENTIONS:
Drug: Chlorhexidine gluconate — Chlorhexidine gluconate (CHG) is a cationic bisguanide that works through disruption of cell membranes. CHG has broad spectrum activity against gram-positive bacteria and to a lesser extent gram negative bacteria. CHG has significant residual activity and addition of alcohol based preparations results in even greater residual activity compared to alcohol alone. CHG acts in the presence of organic material (e.g., blood and biofilm) and its antimicrobial activity is slower than that of alcohols.
  Prevantics® 1 ml Swab contains a cutaneous solution of 3.15% w/v chlorhexidine gluconate (CHG) and 70% v/v isopropyl alcohol (IPA), which is commonly used for the preparation of a patient's skin prior to surgery or venipuncture. Prevantics® Swab is available as a single use pre-moistened 2-sided applicator (1.0 ml).
  Arms: Chlorhexidine Swabs
Drug: Isopropyl Alcohol 70% Topical Application Solution — Isopropyl alcohol (IPA), a topical skin disinfectant, is effective against many pathogens and is commonly supplied as 2x2 inch pre-soaked, single-use gauze wipes.
  Arms: Usual Care
Behavioral: Skin Prep Before Injecting Recreational/Street Drugs — During a single 10 minute session, a healthcare provider gives the participant verbal and written information, counseling, and training to reinforce participant knowledge, motivation, and skills to practice skin swabbing correctly and routinely before injecting.

SUMMARY:
The study examined chlorhexidine gluconate (CHG) swabs as a skin disinfectant in combination with a single-session safer injection training to prevent skin and soft tissue infections (SSTI) in people who inject drugs.

DETAILED DESCRIPTION:
Skin and soft tissue infections (SSTI) are a serious and preventable complication of intravenous drug use, yet few interventions have been developed to reduce SSTI in people who inject drugs (PWID). This study tested two interventions to reduce SSTI in PWID: 1) a single-session behavioral intervention to inculcate skin swabbing behaviors, and 2) chlorhexidine swabs to be used as for cleaning the skin prior to injecting.

ELIGIBILITY:
Inclusion Criteria:

* Self-report intravenous drug use within past 30 days

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Frequency of Skin Swabbing | 2 weeks after randomization
  This question asks how often participants use isopropyl alcohol or chlorhexidine gluconate swabs to disinfect their skin before injecting drugs (never, rarely, occasionally, sometimes, frequently, usually, always)

SECONDARY OUTCOMES:
Swab Acceptability Rating | 2 weeks after randomization
  9-items measure swab acceptability, convenience, safety, ease of use, usefulness, tolerability, satisfaction, and self-efficacy
Safer Injection Knowledge and Behaviors | 2 weeks after randomization
  7-items measure participant knowledge, motivation, and behaviors about skin swabbing to prevent skin and soft tissue infections.

OTHER OUTCOMES:
Skin and Soft Tissue Infection Rate | 2 weeks after randomization
  Assessed as redness, swelling, tenderness at an injection site.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data requests referencing Protocol #2018-0488 should be emailed to Gabriel Culbert (gculbert@uic.edu) and include a statement of how the data will be used and stored.